CLINICAL TRIAL: NCT07349992
Title: Flexible Ureterorenoscopy With High-Power Holmium: YAG Laser and Flexible, Navigable Suction Access Sheath vs Mini-Percutaneous Nephrolithotomy in 2-3 cm Kidney Stones Treatment: A Prospective Cohort Study
Brief Title: Retrograde Intrarenal Surgery (RIRS) With High-Power Laser and Flexible, Navigable Suction Access Sheath (FANS) vs Mini-Percutaneous Nephrolithotomy (miniPCNL) for 2-3 cm Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Muzaffer Tansel Kilinc, MD, Principal Investigator, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIRS-MiniPCNL-2022
Record Dates: First submitted 2026-01-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones; Nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde Intrarenal Surgery (RIRS) Group (Experimental): Intervention: Procedure-Retrograde Intrarenal Surgery
  Interventions: Procedure: Retrograde Intrarenal Surgery
- Mini-Percutaneous Nephrolithotomy (MiniPCNL) Group (Experimental): Intervention: Procedure- Mini Percutaneous Nephrolithotomy
  Interventions: Procedure: Mini Percutaneous Nephrolithotomy

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery — We performed retrograde intrarenal surgery combined with a high-power Holmium:YAG laser and flexible navigable suction access sheath in patients with 2-3 cm renal stones.
  Arms: Retrograde Intrarenal Surgery (RIRS) Group
Procedure: Mini Percutaneous Nephrolithotomy — We performed mini-percutaneous nephrolithotomy in patients with 2-3 cm renal stones.
  Arms: Mini-Percutaneous Nephrolithotomy (MiniPCNL) Group

SUMMARY:
This prospective cohort study aims to compare the safety and efficacy of retrograde intrarenal surgery combined with a high-power Holmium:YAG laser and flexible navigable suction access sheath versus mini-percutaneous nephrolithotomy in patients with 2-3 cm renal stones.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Kidney stones measuring 2-3 cm
* Suitable for Retrograde Intrarenal Surgery (RIRS) or Mini-Percutaneous Nephrolithotomy (MiniPCNL)
* Provided written informed consent

Exclusion Criteria:

* Pregnancy
* Renal transplantation
* Congenital renal anomalies
* Uncorrectable coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Stone-Free Rate | 1 month

SECONDARY OUTCOMES:
Hemoglobin change | postoperative first day
Fluoroscopy time | Perioperative
Complications | up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Medical Faculty, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol